CLINICAL TRIAL: NCT01739166
Title: Child Healthcare Excellence Center - A University-Practice-Public Partnership (CHEC-UPPP)
Brief Title: QI Study of a Practice Facilitator's Impact in Working With Clinics on Improving Dental, Lead & Obesity Measures for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Ohio Department of Job and Family Services (Unknown)
Responsible Party: Principal Investigator, Sharon Meropol, MD, PhD, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10-10-07
Record Dates: First submitted 2012-11-27; First posted 2012-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Lead Poisoning; Obesity; Dental Decay
Keywords: Health Services Research; Quality Assurance
MeSH Terms: conditions — Lead Poisoning; Obesity; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Practice-tailored intervention - Early/Phase 1 (Experimental): During the 6 month Intervention Phase the Practice Facilitator works with each practice to create changes that are tailored to their individual preferences and methods of operation. Sites randomized to Early/Phase 1 start their 6 month intervention immediately after randomization.
  Interventions: Other: Practice-tailored intervention to increase rates of targeted services
- Practice-tailored intervention - Late/Phase 2 (Experimental): The Phase 2 group will start the practice-tailored intervention with the study facilitator 4 months post-randomization and continue through post-randomization month 10.
  Interventions: Other: Practice-tailored intervention to increase rates of targeted services

INTERVENTIONS:
Other: Practice-tailored intervention to increase rates of targeted services — Over a 6 month period, the Practice Facilitator (PF), offers individualized suggestions, strategies and tools for streamlining processes and incorporating new ideas into the flow of a practice's work day to increase their rates of delivery of the 3 targeted services of lead screening, obesity detection and dental decay prevention.
  During the intervention visits the PF reviews a small number of recent well-visit charts. This allows for rapid feedback to a practice on their progress as they work toward reaching outcome measures. It also provides 'real time' feedback regarding the degree to which suggested interventions are working, allowing the PF to change the approach as needed.

SUMMARY:
Funded by the Ohio Department of Job and Family Services - Medicaid Technical Assistance and Policy Program (MEDTAPP), the "Child Health Excellence Center - a University-Practice-Public Partnership" (CHEC-UPPP) focuses on improving the health of Ohio's children in 3 target areas: 1) prevention of dental decay; 2) detection and management of overweight and obesity; and 3) lead screening. These topics represent critical public health issues for Ohio's children.

The study is based on strong evidence that interventions are needed to improve practice in the target areas and that achieving these goals represents fundamental improvements in child health care that would reduce morbidity and costs. The approach for the study involves a trained Practice Facilitator (PF) working with multiple pediatric and family medicine practices to create change tailored to individual practice preferences and methods of operation.

Our overall hypothesis is that a university-community consortium, utilizing evidence-based methods (involving education plus a facilitated, practice-tailored approach) will increase the rates of targeted services in primary care practices.

DETAILED DESCRIPTION:
The research design involves a sample of 30 primary care practices (a combination of pediatric and family medicine) from across Northeast Ohio who have at least a 20% Medicaid patient population. We are using a cross-over study design. After the run-in period during which baseline data is collected via chart review and all practices receive basic education in the 3 focal areas of lead, dental and obesity screening, the practices will be randomly assigned to one of two groups.

The Phase 1 group will receive the practice-tailored intervention with the Practice Facilitator (PF) starting immediately after randomization and continuing for 6 months. The Phase 2 group will start their practice-tailored intervention with the PF 4 months post-randomization and continue through post-randomization month 10.

This design gives us a natural 'control' group (Phase 2 group) for the first four months post-randomization. The Phase 2 group will have had the same Run-in Phase education as the Phase 1 group, but will not be starting the practice-tailored intervention with the study facilitator for 4 months, at which time they will cross-over to their Intervention Phase.

Both Phase 1 and Phase 2 groups will have a 2 month Follow-up Phase after the completion of their 6 month Intervention Phase. During the Follow-up Phase they will strive to continue reaching the outcome measures on their own without the support of the PF. This will give us an opportunity to assess short-term sustainability of the rates of delivery of services achieved during the Intervention Phase.

ELIGIBILITY:
Inclusion Criteria:

* Practice site has 20% or more Medicaid patient population
* Practice is located in Northeast Ohio

Exclusion Criteria:

* Practice has less than 20% Medicaid patient population
* Practice is out of the targeted area

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Lead screening for at-risk 12 and 24 month olds | At baseline, every 2 months during the 6 month Intervention Phase, and after the 2 month Follow-up Phase
  Assessing the rate of lead screening for eligible (i.e., at risk) 12 and 24 month old children is our primary outcome. This is assessed by chart review in the medical record for the index visit.
Identification of BMI percentile and weight diagnosis catergory in 2-17 year olds | At baseline, every 2 months during the 6 month Intervention Phase, and after the 2 month Follow-up Phase
  Assessing the rate of recorded BMI and 2) and rate of accurate recorded weight diagnosis category (underweight < 5th percentile; healthy weight 5th percentile -<85th percentile; overweight 85th percentile - <95th percentile; or obese > 95th percentile) for children 2-17 years of age is our primary outcome. This is assessed by chart review in the medical record for the index visit.
Application of dental fluoride varnish for 12-36 month olds | At baseline, every 2 months during the 6 month Intervention Phase, and after the 2 month Follow-up Phase
  Assessing the rate of dental fluoride varnish application for eligible children 12-36 months of age is our primary outcome. This is assessed by chart review in the medical record for the index visit or within the preceding 6 months.

SECONDARY OUTCOMES:
Rates of elevated lead levels and appropriate follow-up for 12 and 24 months lead screenings | At baseline, every 2 months during the 6 month Intervention and after the 2 month Follow-up Phase
  Our secondary outcome for lead is assessing the rate of rate of elevated lead levels and appropriate follow-up for elevated lead levels per ODH Testing Requirements and Medical Mgmt Recommendations. This is assessed by chart review in the medical record for the index visit for those who had a lead screening at 12 and 24 months.
Rates of appropriate counseling for nutrition & activity and appropriate screening for co-morbidities | At baseline, every 2 months during the 6 month Intervention Phase, and after the 2 month Follow-up Phase
  Our secondary outcome for obesity is assessing the rate of appropriate counseling for nutrition and activity for those in the healthy weight, overweight or obese categories and the rate of appropriate screening for co-morbidities for those in overweight and obese categories. This is assessed by chart review in the medical record for the index visit for those 2-17 years of age.
Rates of oral screening and referral to a dentist for 12-36 month olds | At baseline, every 2 months during the 6 month Intervention Phase, and after the 2 month Follow-up Phase
  Our secondary outcome for dental decay prevention is assessing the rate of oral screening and referral to a dentist by age 12 months or for abnormal oral screenings.

CONTACTS AND LOCATIONS:
Overall Officials: Leona Cuttler, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospital Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Meropol SB, Schiltz NK, Sattar A, Stange KC, Nevar AH, Davey C, Ferretti GA, Howell DE, Strosaker R, Vavrek P, Bader S, Ruhe MC, Cuttler L. Practice-tailored facilitation to improve pediatric preventive care delivery: a randomized trial. Pediatrics. 2014 Jun;133(6):e1664-75. doi: 10.1542/peds.2013-1578. Epub 2014 May 5. PMID 24799539